CLINICAL TRIAL: NCT00187941
Title: Pilot Trial for Implementation of a Medroxyprogesterone(MPA)Pharmacokinetic(PK) Monitoring Strategy in Patients on Mycophenolate Mofetil(MMF)/FK Based Immunosuppression.
Brief Title: MPA PK Monitoring Strategy With MMF/FK Based Immunosuppression
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CEL470
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2012-06-20 (Estimated); Status verified 2012-06

CONDITIONS: Transplantation, Renal; Immunosuppression
Keywords: transplant; renal; Cellcept; therapeutic drug level; MMF; MPA; immunosuppression
MeSH Terms: interventions — Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CellCept (Other): CellCept + Prograf or Neoral + Steroids
  Interventions: Drug: Mycophenolate Mofetil

INTERVENTIONS:
Drug: Mycophenolate Mofetil — Targeted MPA exposure to 30-60 mg/L/h during the first month post-transplant.
  Other Names: CellCept; MMF; RO 70-0003

SUMMARY:
Individuals absorb Cellcept (MMF/Mycophenolate Mofetil) at different rates and it is difficult to determine an individuals level of Mycophenolate Mofetil (MMF, trade name Cellcept)from a single measurement. We will enroll 20 subjects. Plasma samples to be collected pre-MMF dose (trough level) and at 30 and 120 min after the morning dose of MMF.This will be done weekly for the first month and then monthly for the next 6 mths. We hope to use a calculation of the subjects total MMF level during the first month to set a trough target level to use during the next 6 months.

DETAILED DESCRIPTION:
We would use repeated Areas-Under-the-Curve (AUC-a statistical means of summarizing information from a series of measurements on one individual) during the first month post transplant to establish a therapeutic drug exposure for each single patient. We would use the individual trough level from each individual therapeutic AUC for a subsequent individual trough target range. For the purpose of the study, in order to show that by targeting these individualized Mycophenolic Acid (MPA) trough levels we effectively are keeping the patients within a therapeutic drug exposure range, we would continue to obtain abbreviated AUC's at follow up visits. The investigator would be blind to the results of these AUC's after the first month after transplant in order to allow drug exposure targeting only by trough measurements.

From 4 days post transplant, we would draw blood for abbreviated AUC's at 4-5 subsequent clinic visits within a 4 week time frame. We would change the dose based on each AUC to establish an MPA target exposure above 30 mg/L. The individual trough level corresponding to the each patients AUC on target is going to be used for subsequent pk (pharmacokinetic) monitoring. For example if a patient is on 1250 mg bid of Cellcept and we finally obtain an AUC of 40 mg/L/hr and the trough concentration at the time of this pk profile is 2.5 mg/L, we would subsequently target this patient's trough level above 2.5 mg/L. The subsequent AUC's (only needed for the study, not for the final monitoring strategy once established) would serve to confirm that by targeting the trough above 2.5 mg/L the patient effectively stayed within the AUC target range of 30-60 mg/L.

The investigator would be blinded to the follow up AUC's after the first month because the primary objective of the study is to determine if by trough level targeting therapeutic exposure as measured by AUC can be achieved. The investigators would not be blinded though to the initial AUC's which are used to get the patient initially into a therapeutic target window.

We would not consider dose reductions based on elevated trough levels unless toxicities were present. On the other hand we would act on low levels with dose increases in 250 mg bid increments.

For this study we would propose 20 subjects to be enrolled. Each patient would undergo abbreviated pk sampling 4-5 times between week 1 to 4. Subsequently we would do abbreviated AUC's monthly until month 7. We would enroll all patients including those presenting with slow graft function or delayed graft function except for those patients with early technical failure.

Therefore for the study each patient would undergo approximately 12 abbreviated AUC's in the first 7 month's post transplant. Drop out patients will be replaced by new recruits to obtain an evaluable number of patients.

ELIGIBILITY:
Inclusion Criteria:

* Male and female, age 18-80
* On Cellcept (MMF) and Prograf (tacrolimus) based immunosuppression
* Recipient of cadaveric or living donated kidney transplants

Exclusion Criteria:

* Documented non-compliance prior transplant
* Serum albumin <2.5 mg/dl
* Primary non-function
* Not on Prograf
* Pregnant females
* Active serious digestive system disorder

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-08; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Proportion of patients whose measured AUC falls within or outside the therapeutic MPA target range (30-60 mg/L/h) at any given follow up interval, as average over the whole time period. | 7 months
Proportion of patients achieving one or more therapeutic level AUC. | 7 months

SECONDARY OUTCOMES:
Incidence of acute rejection of transplanted kidney | 7 months
Incidence of potentially MPA related toxicities | 7 months
Number of dose changes needed to achieve MPA AUC target within the first month post-transplant | 1 months
Number of dose changes needed to achieve the individualized MPA trough target levels following the first month. | 6 months
To obtain 20 to 25 intraindividual correlation estimates (of one type or another) within each patient: trough vs. AUC. | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Herwig-Ulf Meier-Kriesche, MD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

REFERENCES:
- [Background] Guerra G, Srinivas TR, Schold JD, Eagan AE, Nawrocki, Shaw L, Kaplan B, Womer K, Meier-Kriesche HU. Prospective Blinded Pharmacokinetic Trial to Establish an Individualized MPA Trough Regimen. American Transplant Congress, San Francisco, California